CLINICAL TRIAL: NCT06293196
Title: Effects of Acupoint Massage Around Eyes on Ocular Biological Indexes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20231107
Record Dates: First submitted 2024-02-01; First posted 2024-03-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Investigating the Effects of Periocular Acupressure on Ocular Biological Indicators
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- standard Chinese acupoint eye exercise group (Experimental): The volunteers performed a set of standard Chinese acupoint eye health exercises.
  Interventions: Other: acupressure
- fake acupoint eye exercise group (Experimental): Volunteers performed a group of fake acupoint eye health exercises, the acupoint design in the place without acupoints.
  Interventions: Other: acupressure
- simple eye closure group (No Intervention): The volunteers only closed their eyes and did not perform acupressure.
- simple distance observation group (No Intervention): The volunteers only looked far without acupressure.

INTERVENTIONS:
Other: acupressure — Massage acupoints and non-acupoint areas around the eyes.
  Arms: fake acupoint eye exercise group; standard Chinese acupoint eye exercise group

SUMMARY:
This study aims to investigate whether the acupoint eye exercise could impact the biological parameters of the eye.

ELIGIBILITY:
Inclusion Criteria:

* healthy people of all ages

Exclusion Criteria:

* presence of systemic diseases
* history of other eye diseases, surgeries, and/or medications, as well as eye trauma
* incomplete healing of the surgical site after eye surgery
* consumption of coffee, tea, or vasodilators within 6 hours before the commencement of the test
* exclusion of children, pregnant, and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect of ocular acupoint massage on ocular blood flow. | Ocular blood flow indicators were measured once at pre-intervention, immediately post-intervention, and at 10, 20, and 30 minutes post-intervention.
  Ocular blood flow indicators were obtained using Optical Coherence Tomography (OCT).
The effect of ocular acupoint massage on intraocular pressure. | Intraocular pressure was measured once before the intervention and once immediately after the intervention.
  Intraocular pressure (IOP) of patients was measured and recorded with the ICARE rebound tonometer.
The effect of ocular acupoint massage on the diameter of Schlemm's canal. | Anterior segment imaging was performed once before and once immediately after the intervention to obtain the diameter values of Schlemm's canal.
  Imaging of the nasal and temporal corneoscleral regions of the right eye was performed using swept-source anterior segment optical coherence tomography (SS-AS-OCT). The diameter of Schlemm's canal was measured manually.
The effect of ocular acupoint massage on the area of Schlemm's canal. | Anterior segment imaging was performed once before and once immediately after the intervention to obtain the area values of Schlemm's canal.
  Imaging of the nasal and temporal corneoscleral regions of the right eye was performed using swept-source anterior segment optical coherence tomography (SS-AS-OCT). The area of Schlemm's canal was measured manually.
The effect of ocular acupoint massage on the width of the trabecular meshwork. | Anterior segment imaging was performed once before and once immediately after the intervention to obtain the width values of the trabecular meshwork.
  Imaging of the nasal and temporal corneoscleral regions of the right eye was performed using swept-source anterior segment optical coherence tomography (SS-AS-OCT). The width of the trabecular meshwork was measured manually.
The effect of ocular acupoint massage on the thickness of the trabecular meshwork. | Anterior segment imaging was performed once before and once immediately after the intervention to obtain the thickness values of the trabecular meshwork.
  Imaging of the nasal and temporal corneoscleral regions of the right eye was performed using swept-source anterior segment optical coherence tomography (SS-AS-OCT). The thickness of the trabecular meshwork was measured manually.
The effect of ocular acupoint massage on the tear film. | The Keratograph was performed once before the intervention and once immediately after the intervention.
  The Keratograph was used to dynamically monitor the tear film break-up location and break-up time in a non-contact manner before and after the intervention, with tear meniscus height measured manually.

SECONDARY OUTCOMES:
The effect of ocular acupoint massage on blood pressure. | Blood pressure was measured once before the intervention and once immediately after it.
  Blood pressure was measured using the cuff pressurization method.
The effect of ocular acupoint massage on heart rate. | Heart rate was measured once before the intervention and once immediately after it.
  Heart rate was monitored using the cuff occlusion method.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China